CLINICAL TRIAL: NCT02696551
Title: Impact of Medical Education of Physician Action 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanxi Dayi Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: The IMPACT2 Project
Record Dates: First submitted 2016-02-23; First posted 2016-03-02 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Spondyloarthritis
Keywords: Medical education; Spondyloarthritis; Physician action
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interventional hospital (Experimental): Interventional hospital, which will receive 3-month medical education
  Interventions: Other: Medical education
- Non-interventional hospital (No Intervention): Non-interventional hospital, which will not receive 3-month medical education.

INTERVENTIONS:
Other: Medical education
  Arms: Interventional hospital

SUMMARY:
This is a retrospective and prospective designed study, included hospitals are 1:1 assigned into two groups: ①Interventional hospital, which will receive 3-month medical education; ②Non-interventional hospital, which will not receive 3-month medical education. During 1 month before education, all the electronic records of outpatients and inpatients who visit the included rheumatologists will be collected and the data of test and evaluation results of spondyloarthritis (SpA) patients diagnosed according to new Assessment of Spondylo-Arthritis International Society (ASAS) criteria will be collected from outpatient electronic records and inpatients medical charts; in the 3 months after education, the same data will be collected and compared with the data before education, and the impact of medical education on physician behaviour will be analyzed. Meanwhile, the understanding and acceptance level will be evaluated by the questionnaire, the differences before and after education and the impact of education on physician cognition will be evaluated.

ELIGIBILITY:
Interventional hospital will be selected based on following criteria:

1. having complete outpatients and inpatients electronic records;
2. more than 50% of registrars and/or consultants in the department participated the professional education event;
3. the department head is willing to participate the clinical audit and provide the information from outpatients and inpatients records for data collection;
4. except for rheumatic diseases have been clearly diagnosed.

Non-interventional hospital will be selected based on following criteria:

1. having complete outpatients and inpatients electronic records;
2. no professional education event covered;
3. the department head is willing to participate the clinical audit and provide the information from outpatients and inpatients records for data collection;
4. except for rheumatic diseases have been clearly diagnosed.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Mean of number of positive SpA feature of newly diagnosed patients with inflammatory back pain, before and after the (no-)event | 1 month before (no-) education vs. 3 months after (no-) education
Proportion of patients with a image examination of sacroiliitis ( x-rays, CT, or MRI) in the audit period, before and after the (no-)event | 1 month before (no-) education vs. 3 months after (no-) education
Proportion of patients with a assessment of disease activity in the audit period, before and after the (no-)event | 1 month before (no-) education vs. 3 months after (no-) education

SECONDARY OUTCOMES:
Proportion of patients with a clear diagnosis (Diagnostic for Spondyloarthritis with new ASAS criteria) or receiving a new diagnosis in the audit period, before and after the (no-)event | 1 month before (no-) education vs. 3 months after (no-) education
Mean of the number of physical examinations of disease activity in the audit period, before and after the (no-)event | 1 month before (no-) education vs. 3 months after (no-) education
Change of questionnaire scores of physician in the audit period, before and after the (no-)event | 1 month before (no-) education vs. 3 months after (no-) education
Change of utilization rate of Non Steroidal Anti Inflammatory Drugs (NSAIDs) before and after the (no-)event | 1 month before (no-) education vs. 3 months after (no-) education
Change of utilization rate of biological medication before and after the (no-)event | 1 month before (no-) education vs. 3 months after (no-) education

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Dayi Hospital, Taiyuan, Shanxi, China